CLINICAL TRIAL: NCT03212625
Title: The Effect of Urea Cream on Sorafenib-associated Hand-Foot Skin Reaction in Patients With Korean Hepatocellular Carcinoma Patients: Multicenter, Prospective Randomized Double-Blind Controlled Study
Brief Title: The Effect of Urea Cream on Sorafenib-associated Hand-Foot Skin Reaction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Principal Investigator, Ji Hoon Kim, Associate professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KUGH15337
Record Dates: First submitted 2017-07-02; First posted 2017-07-11 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Urea Cream; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urea cream 20% (Experimental): 144 patients spread urea cream (urea 20%)
  Interventions: Drug: Urea Cream 20%
- Placebo (Placebo Comparator): 144 patients spread placebo cream (urea 0%)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Urea Cream 20% — Sorafenib 400mg (twice daily), Spread urea cream (urea 20%)
  Other Names: Urea group
  Arms: Urea cream 20%
Drug: Placebos — Sorafenib 400mg (twice daily), Spread placebo cream (urea 0%)
  Other Names: Placebo group
  Arms: Placebo

SUMMARY:
Many investigators have studied for prevention and care of Hand-Foot Skin Reaction(HFSR), and urea cream is typical representative. Recent study was performed prevention effect of urea cream for Hand-Foot Skin Reaction(HFSR) on 871 Chinese. But the study did not designed as placebo-control group and it had big defect in double-blinded.

Therefore, it needs complementary study as double-blinded placebo-controlled trial and effect of urea cream on Korean patient group.

DETAILED DESCRIPTION:
Sorafenib is multiple tyrosine kinase inhibitor. It blocks path that such as Raf-1, Vascular Endothelial Growth Factor Receptor (VEGFR), Platelet-Drived Growth Factor Receptor-β (PDGFR-β), c-Jit, Flt-3. Sorafenib was known to increase life rate about processed hepatocellular carcinoma. So it is advised as standard treatment for liver cancer patient who has processed Barcelona Clinic Liver Cancer (BCLC) disease period C.

Sorafenib related side effect has reported such as fatigue, diarrhea, vomit, nausea, pruritus, depilation, Hand-Foot Skin Reaction(HFSR). Among the symptoms, Hand-Foot Skin Reaction(HFSR) is the most occurrence after using sorafenib and major reason of drug dose de-escalation, it function as decrease anti-cancer effect of sorafenib. It is known for the reason of Hand-Foot Skin Reaction(HFSR) occurrence is caused by tyrosine kinase inhibitive action, and its characteristic symptom is known as keratocyte necrosis, dermal edema, parakeratosis, hyperkeratosis. The level is categorized grade 1,2,3 according to the severity.

The result of meta-analysis of 24 clinical trials that contained 6000 patients, Hand-Foot Skin Reaction(HFSR) occured 39% of sorafenib used patients and 9% of total patients had grade 3 Hand-Foot Skin Reaction(HFSR). But prevalence rate on hepatocellular carcinoma patients who used sorafenib is about 51% on Japanese, 45% on Asia-pacific patient (inclusive Korean) and 73.6% on Chinese. Prevalence rate of Hand-Foot Skin Reaction(HFSR) is different from result of each study, but about 50% of sorafenib used patients has had Hand-Foot Skin Reaction(HFSR) generally and Asian has more higher degree of prevalence rate. Therefore, prevent and care of Hand-Foot Skin Reaction(HFSR) on Korean hepatocellular carcinoma patients who used sorafenib is required.

Urea cream is typical representative for prevention and care of Hand-Foot Skin Reaction(HFSR). As stability-guaranteed drug, it is relatively cheap, locally affect and has used for psoriasis treatment. Also it is known for curative effacement on Hand-Foot Skin Reaction(HFSR) after use tyrosine kinase inhibitor such as sorafenib, sunitinib.

Therefore, it needs complementary study as double-blinded placebo-controlled trial and effect of urea cream on Korean patient group.

ELIGIBILITY:
Inclusion Criteria:

* Patient who was diagnosed with hepatocellular carcinoma, and was accompanied by impossible for radical treatment in disease period or do not reaction for local treatment, and the first time for sorafenib injection.
* Standard of hepatocellular carcinoma diagnosis (2014, The Korean Liver Cancer Association)

  1. Suitable on hepatocellular carcinoma pathologically
  2. Hepatic nodule size over 1 cm on high-risk patients(hepatitis B virus positive, hepatitis C virus positive and liver cirrhosis) that identified by ultrasonography : In the case of suitable on hepatocellular carcinoma on over in one or two more dynamic contrast enhanced CT, dynamic contrast enhanced MRI, or MRI with Gadolinium Ethoxybenzyl Diethylenetriamine Pentaacetic Acid(Gd-EOB-DTPA)
  3. Hepatic nodule size under 1 cm on high-risk patients that identified by ultrasonography : serum Alpha-fetoprotein(AFP) elevated over normal range constantly when hepatitis activity was restrained, and the case of suitable on hepatocellular carcinoma on over in two more the above image diagnoses

Exclusion Criteria:

* Unsuitable on inclusion criteria
* Patient who has had systemic anticancer therapy before (including sorafenib)
* Patient who is receiving another treatment to hepatocellular carcinoma recent 3 weeks (allow to local treatment of metastasis lesion only)
* Pregnant or Breastfeeding
* Urea cream contraindication patient (Acute eczema, Inflammatory dermatopathy and Hypersensitivity on Urea and Methylparaben)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of Hand-Foot Skin Reaction(HFSR) on each group | 12 weeks treatment
  Comparison of cumulative incidence of HFSR between placebo group and urea cream group

SECONDARY OUTCOMES:
Cumulative incidence of severe HFSR on each group | 12 weeks treatment
  Comparison of cumulative incidence of severe HFSR (grade 2 or grade 3) between placebo group and urea cream group
Incidence of dose reduction or discontinuation of sorafenib due to HFSR on each group | 12 weeks treatment
  Comparison of incidence of dose reduction or discontinuation of sorafenib due to HFSR on each group
Assessment of Quality Of Life (QOL) | 12 weeks treatment
  Assessment of QOL related to HFSR using The Hand-Foot Skin Reaction and Quality of Life Questionnaire (HF-QoL) scoring system. HF-QOL instrument comprises a 20-item symptom scale and an 18-item daily activity scale. Each item was scored from 0 (not at all) to 4 (always or extremely). Therefore, the range of score for HF-QoL was from 0 to 152 points. (Ref. Anderson et al. The Oncoligist 2015;20:831-838)
Overall survival | 12 weeks treatment
  Overall survival of patients
Tumor response | 12 weeks treatment
  Tumor response using mRECIST criteria
Other side effect | 12 weeks treatment
  The occurrence rate of other side effect excluding HFSR
Incidence of HFSR on 2, 4, 8, and 12 weeks on each group | 2, 4, 8, and 12 weeks
  Comparison of incidence of HFSR on 2, 4, 8, and 12 weeks between placebo group and urea cream group

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hoon Kim, MD, Principal Investigator — Associate Professor
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilhelm SM, Carter C, Tang L, Wilkie D, McNabola A, Rong H, Chen C, Zhang X, Vincent P, McHugh M, Cao Y, Shujath J, Gawlak S, Eveleigh D, Rowley B, Liu L, Adnane L, Lynch M, Auclair D, Taylor I, Gedrich R, Voznesensky A, Riedl B, Post LE, Bollag G, Trail PA. BAY 43-9006 exhibits broad spectrum oral antitumor activity and targets the RAF/MEK/ERK pathway and receptor tyrosine kinases involved in tumor progression and angiogenesis. Cancer Res. 2004 Oct 1;64(19):7099-109. doi: 10.1158/0008-5472.CAN-04-1443. PMID 15466206
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Bruix J, Sherman M; American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma: an update. Hepatology. 2011 Mar;53(3):1020-2. doi: 10.1002/hep.24199. No abstract available. PMID 21374666
- [Background] Chu D, Lacouture ME, Fillos T, Wu S. Risk of hand-foot skin reaction with sorafenib: a systematic review and meta-analysis. Acta Oncol. 2008;47(2):176-86. doi: 10.1080/02841860701765675. PMID 18210295
- [Background] Zhang L, Zhou Q, Ma L, Wu Z, Wang Y. Meta-analysis of dermatological toxicities associated with sorafenib. Clin Exp Dermatol. 2011 Jun;36(4):344-50. doi: 10.1111/j.1365-2230.2011.04060.x. Epub 2011 Apr 20. PMID 21507035
- [Background] Iijima M, Fukino K, Adachi M, Tsukamoto T, Murai M, Naito S, Minami H, Furuse J, Akaza H. Sorafenib-associated hand-foot syndrome in Japanese patients. J Dermatol. 2011 Mar;38(3):261-6. doi: 10.1111/j.1346-8138.2010.01059.x. Epub 2010 Nov 2. PMID 21342228
- [Background] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Background] Ren Z, Zhu K, Kang H, Lu M, Qu Z, Lu L, Song T, Zhou W, Wang H, Yang W, Wang X, Yang Y, Shi L, Bai Y, Guo X, Ye SL. Randomized controlled trial of the prophylactic effect of urea-based cream on sorafenib-associated hand-foot skin reactions in patients with advanced hepatocellular carcinoma. J Clin Oncol. 2015 Mar 10;33(8):894-900. doi: 10.1200/JCO.2013.52.9651. Epub 2015 Feb 9. PMID 25667293
- [Background] Lacouture ME, Wu S, Robert C, Atkins MB, Kong HH, Guitart J, Garbe C, Hauschild A, Puzanov I, Alexandrescu DT, Anderson RT, Wood L, Dutcher JP. Evolving strategies for the management of hand-foot skin reaction associated with the multitargeted kinase inhibitors sorafenib and sunitinib. Oncologist. 2008 Sep;13(9):1001-11. doi: 10.1634/theoncologist.2008-0131. Epub 2008 Sep 8. PMID 18779536
- [Background] Anderson RT, Keating KN, Doll HA, Camacho F. The Hand-Foot Skin Reaction and Quality of Life Questionnaire: An Assessment Tool for Oncology. Oncologist. 2015 Jul;20(7):831-8. doi: 10.1634/theoncologist.2014-0219. Epub 2015 Jun 17. PMID 26084809
- [Derived] Lee YS, Jung YK, Kim JH, Cho SB, Kim DY, Kim MY, Kim HJ, Seo YS, Yoon KT, Hong YM, Lee JH, Lee HW, Yim HJ, Jang BK, Jang ES, Jang JY, Hwang SY. Effect of urea cream on sorafenib-associated hand-foot skin reaction in patients with hepatocellular carcinoma: A multicenter, randomised, double-blind controlled study. Eur J Cancer. 2020 Nov;140:19-27. doi: 10.1016/j.ejca.2020.09.012. Epub 2020 Oct 8. PMID 33039810